CLINICAL TRIAL: NCT03359551
Title: Natural History of the Progression of Choroideremia Study
Acronym: NIGHT
Status: Completed | Type: Observational
Sponsor: NightstaRx Ltd, a Biogen Company (Other)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Other Study IDs: 273CH001; NSR-CHM-OS1 (Other: NightstaRx Ltd, a Biogen Company)
Record Dates: First submitted 2017-11-24; First posted 2017-12-02 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Choroideremia
Keywords: REP1; Retina; Retinal Degeneration; Retinal Dystrophy; Natural History
MeSH Terms: conditions — Choroideremia; Retinal Degeneration; Retinal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this natural history study is to gain a better understanding of the progression of choroideremia (CHM) and add to the knowledge base for this rare disease.

DETAILED DESCRIPTION:
This study was previously posted by NightstaRx Ltd. In October 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Are willing and able to provide informed consent for participation in the study.
* Have a clinical phenotype and confirmed genetic diagnosis of CHM.
* Have active disease clinically visible within the macular region.
* Are willing and able to undergo ophthalmic examinations once every 4 months for up to 20 months.
* Have a BCVA better than or equal to 6/60 (20/200; decimal 0.1; LogMAR 1.0; 34-38 ETDRS letters) in at least one eye.

Key Exclusion Criteria:

* Have a history of amblyopia in the eligible eye.
* Have any other significant ocular or non-ocular disease/disorder in the eligible eye which, in the opinion of the investigator, may put the subject at risk because of participation in the study, influence the results of the study or influence the subject's ability to participate in the study.
* Have participated in an interventional research study in the past 6 months.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) using the Early Treatment Diabetic Retinopathy Study (EDTRS) | Up to Month 20
  BCVA will be assessed for both eyes using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is to be reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.

SECONDARY OUTCOMES:
Change from Baseline in Reading Performance using International Reading Speed Texts (IReST) | Baseline up to Month 12
  Reading performance will be evaluated prior to pupil dilation.
Change from Baseline in Color Vision | Baseline up to Month 12
  Colour vision will be tested prior to pupil dilation. Each eye will be tested separately and in the same order.
Change from Baseline in Visual Fields | Baseline up to Month 12
  The progression of defects in visual fields will be assessed in both eyes using perimetry equipment.
Change from Baseline in Contrast Sensitivity | Baseline up to Month 12
  Contrast sensitivity will be measured for both eyes, prior to pupil dilation, using a Pelli Robson chart.
Change from Baseline in Retinal Thinning Using Spectral Domain Optical Coherence Tomography (SD-OCT) | Baseline up to Month 20
  SD-OCT measurements will be performed after dilation of the participant's pupil.
Change from Baseline in Area of Viable Retinal Tissue Using Fundus Autofluorescence | Baseline up to Month 20
  Fundus Autofluorescence will be performed after dilation of the participant's pupil to assess changes in the area of viable retinal tissue.
Change from Baseline in Retinal Sensitivity Using Microperimetry | Baseline up to Month 20
  Macular analyser integrity assessment (MAIA) microperimetry will be conducted for both eyes to assess changes in retinal sensitivity within the macula.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (20):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Miami, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin
- Research Site, São Paulo, Brazil
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Montreal
  - Research Site, Vancouver
- Research Site, Glostrup Municipality, Denmark
- Research Site, Helsinki, Finland
- Research Site, Montpellier, France
- Germany (2):
  - Research Site, Bonn
  - Research Site, Tübingen
- Research Site, Nijmegen, Netherlands
- United Kingdom (3):
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- [Background] Hariri AH, Velaga SB, Girach A, Ip MS, Le PV, Lam BL, Fischer MD, Sankila EM, Pennesi ME, Holz FG, MacLaren RE, Birch DG, Hoyng CB, MacDonald IM, Black GC, Tsang SH, Bressler NM, Larsen M, Gorin MB, Webster AR, Sadda SR; Natural History of the Progression of Choroideremia (NIGHT) Study Group. Measurement and Reproducibility of Preserved Ellipsoid Zone Area and Preserved Retinal Pigment Epithelium Area in Eyes With Choroideremia. Am J Ophthalmol. 2017 Jul;179:110-117. doi: 10.1016/j.ajo.2017.05.002. Epub 2017 May 10. PMID 28499705